CLINICAL TRIAL: NCT06068777
Title: Scentsational Smiles: The Impact of Aromatherapy on Alleviating Dental Anxiety in Children
Brief Title: The Impact of Aromatherapy on Alleviating Dental Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 455/2022
Record Dates: First submitted 2023-07-08; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Pain Syndrome
MeSH Terms: conditions — Somatoform Disorders | interventions — lemongrass oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): with no interference before dental anesthesia and extraction
- Rosemary group (Active Comparator): children inhaled two drops of rosemary oil for 3 minutes before the procedures of dental anesthesia and extraction of a primary molar,
  Interventions: Drug: Rosmary
- Lemongrass group (Active Comparator): children inhaled two drops of lemongrass oil, for 3 minutes before the procedure of dental anesthesia and extraction of a primary molar
  Interventions: Drug: Lemongrass Oil

INTERVENTIONS:
Drug: Rosmary — inhale two drops of rosemary oil, from a gauze, for 3 minutes before the procedure of extraction of a primary molar
  Arms: Rosemary group
Drug: Lemongrass Oil — inhale two drops of lemongrass oil, from a gauze, for three minutes before the procedure of extraction.
  Arms: Lemongrass group

SUMMARY:
Dealing with dental anxiety in children is the most problematic responsibilities for pedodontists in the dental office. Essential oils had been used for reducing dental anxiety in adults; this study is a challenge to understand their effects on children. Aromatherapy is considered as a reasonable, potent, safe, and non-pharmacological way, which has been taken into consideration, especially for children who are supposed to go through any dental procedure under local anesthesia. The aim of this study is to explore and compare the effect of Rosemary versus Lemongrass essential oils on dental anxiety levels and vital signs of children during dental anesthesia and extraction of a lower primary molar in a dental office. Forty-five children, aged between 4 to 7 years, who had a minimum of one mandibular primary molar with deep caries indicated for extraction were selected. Patients are divided, randomly, into three groups (15 children each): Group I (control group): with no interference before dental anesthesia and extraction, Group II (Rosemary group): children inhaled two drops of rosemary oil for 3 minutes before the procedures of dental anesthesia and extraction of a primary molar, Group III (Lemongrass group): children inhaled two drops of lemongrass oil, for 3 minutes before the procedure of dental anesthesia and extraction of a primary molar. Wong Baker Scale and the physiological measures of the children's anxiety will be evaluated and recorded for each child by measuring (pulse rate, oxygen saturation, and blood pressure) before, during and after the dental procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from six to nine years old
* Both girls and boys will be included.
* Patients who need extraction in at least one primary molar.
* Parents who will agree to contribute in the study.
* Patients with Frankl Behavior Rating Scale, categories 2, 3 and 4

Exclusion Criteria:

* Medically compromised patient
* Allergic children

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
measuring pulse rate " heart rate" | baseline before procedure, during procedure "extraction" and immediately after procedure "extraction"
oxygen saturation | baseline before procedure, during procedure "extraction" and immediately after procedure "extraction"
  oxygen saturation using pulse oximeter.
blood pressure using a sphygmomanometer | baseline before procedure, during procedure "extraction" and immediately after procedure "extraction"
  systolic and diastolic blood pressure will be measured
pain level | baseline before procedure, during procedure "extraction" and immediately after procedure "extraction"
  the Wong-Baker Scale will be used where 0 no pain and 7 hurts worst

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No